CLINICAL TRIAL: NCT00050856
Title: Multicenter, Open-Label, Early Acces Program of Fuzeon (Enfuvirtide T-20/Ro 29,9800, HIV-1 Fusion Inhibitor) in Combination With Free Choice Antiretroviral Regimen to Assess Serious Adverse Events, Serious AIDS-Defining Events, and Tolerability in Patient
Brief Title: Fuzeon (Enfuvirtide) Early Access Program for Patients With HIV-1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030056; 03-I-0056
Record Dates: First submitted 2002-12-23; First posted 2002-12-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-11

CONDITIONS: HIV Infections
Keywords: Antiretrovial Therapy; Salvage; CD4+Lymphocyte Count; HIV-1 RNA Level; Subcutaneous Injection
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Enfuvirtide T/20/Ro 29,9800, HIV-1 Infusion Inhibitor

SUMMARY:
This study will determine the safety and tolerability of Fuzeon (enfuvirtide) used together with other treatments for HIV infection in patients with advanced HIV disease. Fuzeon is an antiretroviral drug. Unlike other antiretrovirals, however, which work against the virus once it is already in the cell, Fuzeon prevents the virus from getting into healthy cells.

Patients 18 years of age and older with advanced HIV-1 infection, who do not respond to approved antiretroviral therapy, may be eligible for this study. Candidates must have a CD4 lymphocyte count less than 100 cells/mm3 and a viral load greater than 10,000 copies/mL. They will be screened with a medical history, physical examination, and blood tests, and may also have an electrocardiogram (ECG), chest x-ray and urine test.

Patients enrolled in the study will be re-examined and have additional blood tests before beginning treatment with Fuzeon. They will then be taught how to self-inject the medicine under the skin and will take two doses daily (less than 1/4 teaspoon each), 12 hours apart. After the first treatment, participants will have follow-up visits at weeks 1, 2, 4, 8, 12, 24, 36, 48, and every 12 weeks after that, if necessary, until 12 weeks after the drug becomes commercially available. Visits may be scheduled more often if a problem arises. During the follow-up visits, patients will have blood drawn, and their blood pressure, pulse rate and temperature will be checked. They will also report any drug side effects they have experienced.

Patients may continue to take Fuzeon as long as they benefit from therapy and do not experience severe side effects from the treatment. The drug will be provided to participants until 12 weeks after it is sold in the United States.

DETAILED DESCRIPTION:
Over the last few years, an unprecedented decrease in the mortality and morbidity associated with AIDS has been achieved attributed to the use of highly active antiretroviral therapy (HAART) which consists of three different classes of drugs: Nucleoside reverse transcriptase inhibitors (NRTIs), protease inhibitors (PIs), and non-nucleoside reverse transcriptase inhibitors (NNRTIs). However, the durability of viral suppression is often limited by treatment with combinations of non-fully suppressive antiretroviral agents. Heavily pretreated patients often possess multiple mutations of the reverse transcriptase and protease genes resulting in multi-drug resistance. Thus, a pharmacological agent effective at an alternate point in the virus replication cycle would make a valuable addition to the anti-HIV armamentarium. T-20, enfuvirtide, is the first drug to be developed which specifically inhibits the function of the gp41 transmembrane glycoprotein of HIV-1. The objective of this study is to assess the safety and tolerability of Fuzeon (Enfuvirtide) in patients who are limited by the current commercially available antiretroviral agents or agents available via early access or compassionate use programs as per the judgment of the investigator or patients with advanced disease and most in need of therapy. This study is a multicenter, open-label, single-arm, safety study. Each patient will receive enfuvirtide 90 mg (deliverable dose) via subcutaneous injection twice daily with food, in combination additional antiretroviral agents. Subjects will continue to receive enfuvirtide until 12 weeks after commercial availability of enfuvirtide in the United States. Laboratory testing, CD4+lymphocyte counts, HIV-1 viral loads will be monitored on a regular and continual basis. The main outcome measures are ones of safety and tolerability: serious adverse events (including all deaths, serious AIDS defining events, and discontinuations for any reason), injection reconstitution fatigue.

ELIGIBILITY:
INCLUSION CRITERIA:

To be eligible for this trial, patients must fulfill all inclusion criteria listed below:

1. Male and female HIV-1 infected adults or adolescents (greater than or equal to 16 years of age).
2. CD4 lymphocyte count less than or equal to 100 cells/mm(3) and HIV-1 RNA viral load greater than or equal to 10,000 copies/mL while on HAART (latest available measurement must be within the last 90 days).
3. Patients must be limited by the current commercially available antiretroviral agents or agents available via Early Access or Compassionate Use Programs as per the judgment of the investigator OR patients with advanced disease and most in need defined as prior documented drug resistance or have documented evidence of greater than 6 months prior experience to each of the three classes of ARV's.
4. Patients must be able and willing to provide written informed consent (for patients less than 18 years of age, a parent or legal guardian must also sign the Informed Consent Form).
5. Women of childbearing potential must have a documented negative pregnancy test at baseline and ensure that two reliable forms of contraception are being used, including a barrier method, for the duration of the study, and for 90 days after the last dose of study medication.

EXCLUSION CRITERIA:

Patients meeting any of the following exclusion criteria will not be eligible for participation in this trial:

1. Female patients who are pregnant, breast-feeding, or who plan to become pregnant or breast-feed during the study.
2. Any current clinical or laboratory parameter of ACTG grade 4. Asymptomatic grade 4 abnormalities will be permitted, at the discretion of the investigator, if the potential benefit of treatment outweighs the potential risk.
3. Evidence of ongoing alcohol and/or drug or substance abuse that, in the judgment of the investigator, would result in the patient being unreliable in fulfilling the conditions of this protocol.
4. Prior non-adherence to antiretroviral treatment regimens that, in the judgment of the investigator, resulted in the patient's failing prior regimens and which would likely result in the patient being unreliable in fulfilling the conditions of this protocol.
5. Inability to self-inject Fuzeon (enfuvirtide) as indicated in the protocol, unless a reliable caregiver is willing, able, and available to provide this service on a continuous basis for the duration of the study.
6. Evidence of active, untreated opportunistic infection, intercurrent illness, drug toxicity or any other condition such that, in the judgment of the investigator, the patient would not be able to continue or take a prescribed antiretroviral regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 2002-11; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Mitsuya H, Yarchoan R, Broder S. Molecular targets for AIDS therapy. Science. 1990 Sep 28;249(4976):1533-44. doi: 10.1126/science.1699273.
- [Background] Durant J, Clevenbergh P, Halfon P, Delgiudice P, Porsin S, Simonet P, Montagne N, Boucher CA, Schapiro JM, Dellamonica P. Drug-resistance genotyping in HIV-1 therapy: the VIRADAPT randomised controlled trial. Lancet. 1999 Jun 26;353(9171):2195-9. doi: 10.1016/s0140-6736(98)12291-2. PMID 10392984